CLINICAL TRIAL: NCT02727348
Title: Haemodynamic and Pain Outcomes in Patients Undergoing Diabetic Foot Surgery Performed Under Sciatic Nerve Blocks With or Without Femoral Nerve Block Versus Spinal Anaesthesia
Brief Title: Sciatic Nerve Blocks With or Without Femoral Block Versus Spinal Anaesthesia in Patients Undergoing Diabetic Foot Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Malaya (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 201401-0658
Record Dates: First submitted 2014-04-30; First posted 2016-04-04 (Estimated); Last update posted 2016-04-04 (Estimated); Status verified 2016-03

CONDITIONS: Diabetic Foot
Keywords: femoral sciatic block spinal diabetic foot haemodynamic pain
MeSH Terms: conditions — Diabetic Foot | interventions — Anesthesia, Spinal

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: No

ARMS (2):
- Sciatic block with or without femoral block (Experimental): Sciatic block with or without femoral block performed on the patient with 3mg/kg of ropivacaine
  Interventions: Procedure: Sciatic with or without femoral block
- Spinal anaesthesia (Active Comparator): Spinal anaesthesia will be performed on the patient with heavy marcaine 0.5% up to 3mls
  Interventions: Procedure: Spinal anaesthesia

INTERVENTIONS:
Procedure: Sciatic with or without femoral block — Sciatic with or without femoral block performed either with ultrasound and/or nerve stimulator on the patient with 3mg/kg of ropivacaine
  Arms: Sciatic block with or without femoral block
Procedure: Spinal anaesthesia — Spinal anaesthesia with up to 3mls of 0.5% bupivacaine
  Arms: Spinal anaesthesia

SUMMARY:
Background:

Dysautonomia refers to the abnormal function of the autonomic nervous system including sympathetic and parasympathetic nervous system. Diabetes mellitus causes secondary dysautonomias (1). The Survey of Autonomic Symptoms (SAS) is a simple and validated tool to assess the presence and severity of autonomic symptoms (2).

Diabetic patients also suffer from chronic neuropathic pain. After amputation surgeries, up to 78% of these patients may develop post surgical neuropathic pain (3). The self-report version of the Leeds Assessment of Neuropathic Symptoms and Signs pain scale (S-LANSS) is validated as a diagnostic tool to assess patients with neuropathic pain (4). This scale will be used to assess if there is any changes in the pain experienced after diabetic foot surgery.

Currently, both spinal anaesthesia (SAB) and ultrasound guided femoral and sciatic peripheral nerve blocks (FSNB) are acceptable anaesthesia for dysautonomic diabetic patients with diabetic foot ulcer going for wound debridement, Ray's amputation and below knee amputation (5)

Many studies have compared multiple perioperative parameters of patients undergoing lower limb surgery under peripheral nerve blocks versus spinal anaesthesia. These parameters include preparation time, anaesthetic complications (e.g. hypotension, nausea and vomiting, post-dural puncture headache, urinary retention), patient satisfaction and postoperative pain control (6,7,8).

The investigators want to study if patients with dysautonomia have a different haemodynamic response to spinal anaesthesia or peripheral nerve blockade changes compared to patients with normal autonomic function.

Secondarily, the investigators would also study if there is a difference in post operative pain control as well as incidence in chronic pain in patients who receive spinal anaesthesia versus peripheral nerve blockade.

DETAILED DESCRIPTION:
Dysautonomia refers to the abnormal function of the autonomic nervous system including sympathetic and parasympathetic nervous system. Diabetes mellitus causes secondary dysautonomias (1). The Survey of Autonomic Symptoms (SAS) is a simple and validated tool to assess the presence and severity of autonomic symptoms (2).

Diabetic patients also suffer from chronic neuropathic pain. After amputation surgeries, up to 78% of these patients may develop post surgical neuropathic pain (3). The self-report version of the Leeds Assessment of Neuropathic Symptoms and Signs pain scale (S-LANSS) is validated as a diagnostic tool to assess patients with neuropathic pain (4). This scale will be used to assess if there is any changes in the pain experienced after diabetic foot surgery.

Currently, both spinal anaesthesia (SAB) and ultrasound guided femoral and/or sciatic peripheral nerve blocks (FSNB) are acceptable anaesthesia for dysautonomic diabetic patients with diabetic foot ulcer going for wound debridement, Ray's amputation and below knee amputation (5)

Many studies have compared multiple perioperative parameters of patients undergoing lower limb surgery under peripheral nerve blocks versus spinal anaesthesia. These parameters include preparation time, anaesthetic complications (e.g. hypotension, nausea and vomiting, post-dural puncture headache, urinary retention), patient satisfaction and postoperative pain control (6,7,8).

The investigators want to study if patients with dysautonomia have a different haemodynamic response to spinal anaesthesia or peripheral nerve blockade changes compared to patients with normal autonomic function.

Secondarily, the investigators would also study if there is a difference in post operative pain control as well as incidence in chronic pain in patients who receive spinal anaesthesia versus peripheral nerve blockade.

ELIGIBILITY:
Inclusion Criteria:

* Diabetic patients with diabetic foot ulcer undergoing diabetic foot surgery below the knee

Exclusion Criteria:

* Refuse spinal or regional anaesthesia
* Uncooperative patients
* Patients with contraindication for FSNB or SAB
* Patients with known allergy to local anaesthetics

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2014-05; Primary Completion 2016-01 (Actual); Study Completion 2016-02 (Actual)

PRIMARY OUTCOMES:
Blood pressure or heart rate changes more than 30% of baseline after spinal or block is considered significant | 60 minutes
  haemodymic checks were performed at intervals up to 60 minutes after block or spinal

SECONDARY OUTCOMES:
S-LANSS score in who receive FSNB versus SAB. | 3 months
  S-LANSS score were obtained at 1 day and 3 months after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Chew Yin Wang, MBChB, Study Director — University of Malaya; Hou Yee Lai, MBBS, Principal Investigator — University of Malaya
Locations (1):
- University Malaya Medical Centre, Kuala Lumpur, Kuala Lumpur, Malaysia

REFERENCES:
- [Derived] Lai HY, Foo LL, Lim SM, Yong CF, Loh PS, Chaw SH, Hasan MS, Wang CY. The hemodynamic and pain impact of peripheral nerve block versus spinal anesthesia in diabetic patients undergoing diabetic foot surgery. Clin Auton Res. 2020 Feb;30(1):53-60. doi: 10.1007/s10286-017-0485-8. Epub 2017 Dec 1. PMID 29196938